CLINICAL TRIAL: NCT00946192
Title: Fat Mediated Modulation of Reproductive and Endocrine Function in Young Athletes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Madhusmita Misra, Associate Professor of Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000353; R01HD060827-01A1 (NIH)
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2020-03-18 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Exercise-related Amenorrhea
Keywords: Amenorrhea; Adolescent; Endurance; Athletes; Females; Osteopenia; Osteoporosis; Estrogen
MeSH Terms: conditions — Amenorrhea; Bone Diseases, Metabolic; Osteoporosis | interventions — Progesterone; Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Estrogen Patch (Experimental): 17Beta-estradiol transdermal patch twice weekly application for 12 months
  Interventions: Drug: Transdermal 17Beta-estradiol, progesterone
- Estrogen Pill (Active Comparator): One pill containing estrogen and progesterone taken daily for 21 days followed by placebo pills only for 7 days; regimen repeated for 12 months.
  Interventions: Drug: Ethinyl Estradiol + Desogestrel
- Control (Sham Comparator): Elemental calcium 1200 mg and Vit D 400 IU taken orally daily
  Interventions: Dietary Supplement: Sham Comparator

INTERVENTIONS:
Drug: Transdermal 17Beta-estradiol, progesterone — 100 mcg/day 17Beta-estradiol; transdermal twice weekly application for 12 months (with cyclic micronized progesterone pills (Prometrium): 200 mg taken orally daily Day 1 to Day 12 each month) + Elemental calcium 1200 mg and Vit D 400 IU taken orally daily
  Other Names: Vivelle Dot transdermal patch; Prometrium
  Arms: Estrogen Patch
Drug: Ethinyl Estradiol + Desogestrel — Oral ethinyl estradiol (0.03 mg) + desogestrel (0.15 mg) + Elemental calcium 1200 mg and Vit D 400 IU taken once daily
  Other Names: Apri
  Arms: Estrogen Pill
Dietary Supplement: Sham Comparator — Elemental calcium 1200 mg and Vit D 400 IU taken orally daily
  Arms: Control

SUMMARY:
One aim of this study is to determine changes in body composition and hormones that differentiate athletes who stop getting their periods versus those who continue to get their periods and non-athletes. The second aim of this study is to determine whether transdermal or oral estrogen (versus no estrogen) is effective in increasing bone density and improving bone microarchitecture in adolescent athletes who are not getting their periods and are thus estrogen deficient. The investigators hypothesize that transdermal estrogen will be more effective than oral estrogen or no estrogen in improving bone health in amenorrheic adolescent athletes.

DETAILED DESCRIPTION:
As many as 25% of adolescent and young adult endurance athletes develop amenorrhea, and factors that cause amenorrhea to occur in some, but not all, athletes have not been well characterized. Recent data indicate the critical importance of a negative energy balance state and leptin in regulating the Hypothalamic-pituitary-gonadal (H-P-G) axis. However, these factors do not completely account for alterations in this axis, and other contributing factors are unclear. Our preliminary data indicate the importance of low fat mass and fat related hormones in mediating hypogonadism in young athletes. This study will confirm these data and determine whether low fat mass and altered levels of adipokines, such as leptin and adiponectin, and hormones regulated by fat mass, such as ghrelin and peptide YY (PYY), determine alterations in LH pulsatility. A very concerning impact of amenorrhea in athletes is low bone mineral density (BMD). Preliminary data indicate lower BMD in adolescent athletes with amenorrhea (AA) compared with eumenorrheic athletes (EA) and non-athletic controls. The high prevalence of AA in adolescents is particularly concerning, because this population is potentially at greater risk as it is actively accruing bone. Of importance, bone microarchitecture, a better predictor of bone strength than BMD, has not been studied in AA. Because pubertal increases in estrogen are integral to optimizing peak bone mass, and AA is characterized by hypoestrogenism, this randomized study of transdermal estrogen versus oral estrogen or no estrogen will also examine whether estrogen replacement increases BMD and improves bone microarchitecture in adolescent AA 14-21 years old. EA and sedentary controls will be followed without intervention for this period. Despite the prevalent practice of prescribing oral contraceptives in AA, there is a paucity of data regarding benefits of this intervention in teenagers. Because transdermal estrogen, unlike oral estrogen, does not suppress IGF-1, an important bone anabolic factor, we expect effects of transdermal estrogen to exceed those of oral estrogen or no therapy. In addition, preliminary data indicate that low fat mass and alterations in fat related hormones may contribute to decreased bone accrual rates in athletes, and will be confirmed in this study. To summarize, a better understanding of the pathophysiology of reproductive dysfunction is critical to develop therapeutic strategies that will normalize the reproductive axis and bone accrual, and these are the questions that this study aims to answer.

ELIGIBILITY:
Inclusion Criteria:

* Females 14-21 years old Note: Our pilot data are reassuring in that young women 18-25 years old with hypothalamic amenorrhea are not adversely affected with estrogen use. In fact, in our prospective study, beneficial effects were observed both in young women 18-25 years old using oral estrogen, and in 14-18 year old adolescent girls using transdermal estrogen. We therefore feel that including girls in the 14-21 year age range will not be hazardous to their bone health. In fact, given the lack of data in this age group, it is important to study younger women and teenagers rather than extrapolate data from studies in adults to this younger population. Hormone dynamics differ in teenagers compared with adults, and bone mass accrual is even more dependent on estrogen and IGF-1 in younger than older women who have already achieved peak bone mass.
* Bone age (BA) >15 years Note: 99% of adult height is achieved at a BA of 15 years, thus estrogen replacement will not result in stunting of height potential after this age. Although we could have chosen to include girls with a BA >14 in this study, we are limiting this to girls with a BA of >15 years. This is because 2% of growth potential persists at a BA of 14 years, versus only 1% at a BA of 15 years (~0.6" of potential height (130)). Thus, to avoid potential stunting of growth potential with estrogen replacement, we have chosen to include girls with BA of > 15 years.
* BMI between 10th-90th percentiles for age.
* Amenorrhea (for AA): absence of menses for > three months (74) within a period of oligomenorrhea (cycle length > six weeks) for >six months, or absence of menarche at >16 years.
* Eumenorrhea (EA and controls): > nine menses (cycle length 21-35 days) in preceding year.
* Non-athlete healthy controls will be eligible if weight bearing exercise activity is less than two hours a week and if they are not participating in organized team sports.
* Endurance athletes Note: severity of low BMD and menstrual dysfunction differ by kind of exercise and activity. For example, runners have a higher prevalence of menstrual irregularity than swimmers and cyclists (131). By limiting enrollment to endurance athletes, we will eliminate variability from the type of activity. Endurance training is defined as > 4 h of aerobic weight-bearing training of the legs or specific endurance training weekly, or > 20 miles of running weekly for a period of > 6 months in the last year.

Exclusion Criteria:

* Other conditions that may affect bone metabolism

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusmita Misra, MD, MPH, Principal Investigator — Massachusetts General Hospital Pediatric Neuroendocrine Unit and Harvard Medical School
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ackerman KE, Singhal V, Slattery M, Eddy KT, Bouxsein ML, Lee H, Klibanski A, Misra M. Effects of Estrogen Replacement on Bone Geometry and Microarchitecture in Adolescent and Young Adult Oligoamenorrheic Athletes: A Randomized Trial. J Bone Miner Res. 2020 Feb;35(2):248-260. doi: 10.1002/jbmr.3887. Epub 2019 Nov 7. PMID 31603998
- [Derived] Plessow F, Singhal V, Toth AT, Micali N, Eddy KT, Misra M. Estrogen administration improves the trajectory of eating disorder pathology in oligo-amenorrheic athletes: A randomized controlled trial. Psychoneuroendocrinology. 2019 Apr;102:273-280. doi: 10.1016/j.psyneuen.2018.11.013. Epub 2018 Nov 16. PMID 30639922
- [Derived] Singhal V, Ackerman KE, Bose A, Flores LPT, Lee H, Misra M. Impact of Route of Estrogen Administration on Bone Turnover Markers in Oligoamenorrheic Athletes and Its Mediators. J Clin Endocrinol Metab. 2019 May 1;104(5):1449-1458. doi: 10.1210/jc.2018-02143. PMID 30476179
- [Derived] Ackerman KE, Singhal V, Baskaran C, Slattery M, Campoverde Reyes KJ, Toth A, Eddy KT, Bouxsein ML, Lee H, Klibanski A, Misra M. Oestrogen replacement improves bone mineral density in oligo-amenorrhoeic athletes: a randomised clinical trial. Br J Sports Med. 2019 Feb;53(4):229-236. doi: 10.1136/bjsports-2018-099723. Epub 2018 Oct 9. PMID 30301734
- [Derived] Baskaran C, Cunningham B, Plessow F, Singhal V, Woolley R, Ackerman KE, Slattery M, Lee H, Lawson EA, Eddy K, Misra M. Estrogen Replacement Improves Verbal Memory and Executive Control in Oligomenorrheic/Amenorrheic Athletes in a Randomized Controlled Trial. J Clin Psychiatry. 2017 May;78(5):e490-e497. doi: 10.4088/JCP.15m10544. PMID 28297591
- [Derived] Ackerman KE, Slusarz K, Guereca G, Pierce L, Slattery M, Mendes N, Herzog DB, Misra M. Higher ghrelin and lower leptin secretion are associated with lower LH secretion in young amenorrheic athletes compared with eumenorrheic athletes and controls. Am J Physiol Endocrinol Metab. 2012 Apr 1;302(7):E800-6. doi: 10.1152/ajpendo.00598.2011. Epub 2012 Jan 17. PMID 22252944
- [Derived] Ackerman KE, Nazem T, Chapko D, Russell M, Mendes N, Taylor AP, Bouxsein ML, Misra M. Bone microarchitecture is impaired in adolescent amenorrheic athletes compared with eumenorrheic athletes and nonathletic controls. J Clin Endocrinol Metab. 2011 Oct;96(10):3123-33. doi: 10.1210/jc.2011-1614. Epub 2011 Aug 3. PMID 21816790

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Estrogen Patch | Estrogen Pill | Control
Started | 43 | 40 | 38
Completed | 25 | 22 | 26
Not Completed | 18 | 18 | 12
Not completed — Lost to Follow-up | 6 | 11 | 9
Not completed — Withdrawal by Subject | 10 | 7 | 3
Not completed — Did not start medication | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Athletes with amenorrhea
Groups:
- Total: Total of all reporting groups
Arm/Group | Estrogen Patch | Estrogen Pill | Control | Total
Number analyzed (Participants) | 43 | 40 | 38 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.86 (0.40) | 20.30 (0.44) | 19.35 (0.38) | 19.84 (0.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 40 | 38 | 121
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 43 | 40 | 36 | 119
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 4 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 37 | 38 | 35 | 110
  More than one race | 1 | 2 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 40 | 38 | 121
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.45 (0.35) | 20.80 (0.39) | 20.75 (0.34) | 20.67 (0.36)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Bone Mineral Density
Description: Change in bone density with transdermal estrogen versus oral estrogen or no estrogen in amenorrheic athletes
Time Frame: 12 months
Measure: Mean (Standard Error); unit: g/cm^2
Arm/Group | Estrogen Patch | Estrogen Pill | Control
Number analyzed (Participants) | 25 | 22 | 26
g/cm^2 | 0.025 (0.011) | 0.008 (0.011) | 0.012 (0.012)
Statistical Analysis 1: Comparison: Estrogen Patch vs Estrogen Pill vs Control; Test type: Other — Least square means; p = 0.039, Mixed Models Analysis

2. Secondary Outcome: Change in Total Volumetric Bone Mineral Density (Tibia)
Description: Change in total volumetric bone density at the tibia with transdermal estrogen versus oral estrogen or no estrogen in amenorrheic athletes
Time Frame: 12 months
Measure: Mean (Standard Error); unit: mg HA/cm^3
Arm/Group | Estrogen Patch | Estrogen Pill | Control
Number analyzed (Participants) | 24 | 24 | 27
mg HA/cm^3 | 7.01 (3.06) | 1.17 (3.05) | 3.71 (4.44)
Statistical Analysis 1: Comparison: Estrogen Patch vs Estrogen Pill vs Control; Test type: Other; p = 0.018, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Estrogen Patch | Estrogen Pill | Control
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 3/43 | 0/40 | 1/38
Other Adverse Events (participants affected / at risk) | 10/43 | 13/40 | 1/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Patch (N=43) | Estrogen Pill (N=40) | Control (N=38)
Fractures or sprains (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Sinus surgery (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estrogen Patch (N=43) | Estrogen Pill (N=40) | Control (N=38)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Dizziness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Breast tenderness (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (General disorders) | 2 (2) | 0 (0) | 0 (0)
Early menses (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Yeast infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Worsening depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Mood swings (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Generalized discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vasovagal response (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased libido (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mononucleosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Skin tags (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte changes (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT00946192/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/92/NCT00946192/SAP_001.pdf